CLINICAL TRIAL: NCT03814356
Title: Stimulant Therapy Targeted to Individualized Connectivity Maps to Promote ReACTivation of Consciousness - A Phase 1 Study
Brief Title: Stimulant Therapy Targeted to Individualized Connectivity Maps to Promote ReACTivation of Consciousness
Acronym: STIMPACT
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Brian L. Edlow, M.D., Director, Laboratory for NeuroImaging of Coma and Consciousness (NICC), Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 140675; DP2HD101400 (NIH)
Record Dates: First submitted 2019-01-15; First posted 2019-01-24 (Actual); Results first posted 2025-10-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Brain Injury Traumatic Severe (Diagnosis); Coma; Consciousness, Level Altered; Anoxic Brain Injury
MeSH Terms: conditions — Disease; Coma; Consciousness Disorders; Hypoxia-Ischemia, Brain | interventions — Methylphenidate; 5,10-dihydro-5-methylphenazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IV MPH (Experimental): All patients will receive IV Methylphenidate (MPH). Patients will receive escalating daily doses of IV MPH starting at 0.5 mg/kg, increasing stepwise to 1.0mg/kg and 2.0 mg/kg unless an adverse event (AE) necessitates dose de-escalation or a serious adverse event (SAE) necessitates that the patient stop participation in the study.
  Interventions: Drug: Methylphenidate

INTERVENTIONS:
Drug: Methylphenidate — IV MPH
  Other Names: MPH

SUMMARY:
Phase 1 of the STIMPACT trial is an open label,dose-escalation,safety study of intravenous (IV) methylphenidate (MPH) therapy in patients with disorders of consciousness (DoC) caused by severe brain injuries.

DETAILED DESCRIPTION:
To be classified as having a DoC, a patient must be in a coma, vegetative state (VS), or minimally conscious state (MCS), as determined by behavioral assessment using the Coma Recovery Scale-Revised (CRS-R). Patients with DoC admitted to the intensive care unit (ICU) will be eligible for the study. A total of 10 patients with DoC will be enrolled in the Phase 1 study. Patients will receive escalating daily doses of IV MPH starting at 0.5 mg/kg, increasing stepwise to 1.0mg/kg and 2.0 mg/kg unless an adverse event (AE) necessitates dose de-escalation or a serious adverse event (SAE) necessitates that the patient stop participation in the study. Pharmacokinetics will be evaluated in selected patients with indwelling venous catheters or arterial catheters via serial serum measurements of MPH at each dose. The pharmacodynamic properties of IV MPH at each dose will be assessed by comparison of pre-versus post-dose EEG-based measures. The pharmacodynamic properties of the maximum tolerated dose will also be assessed by comparison of pre-versus post-dose resting state functional MRI (rs-fMRI) connectivity measures. Finally, we will test the association between structural connectivity of the ventral tegmental area (VTA), a dopaminergic brainstem nucleus that is believed to mediate MPH activation of the cerebral cortex, and EEG and rs-fMRI pharmacodynamic measures.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Severe, acute traumatic brain injury
3. Diagnosis of Coma, Vegetative State, or Minimally Conscious State

Exclusion Criteria:

1. Penetrating brain injury caused by a metallic missile/object (e.g. bullet)
2. Body metal contraindicating MRI
3. Prisoner or ward of the state
4. Neurological

   1. Bilateral dilated unresponsive pupils
   2. Intracranial hypertension (Intracranial Pressure [ICP] > 25 mmHg for > 5 min within past 24 hours with head-of-bed at standard clinical angle of 30-45 degrees)
   3. Intracranial bolt
   4. Status epilepticus or concern for post-ictal state
5. Cardiovascular

   1. Poorly controlled hypertension (SBP > 200 mmHg of DBP > 120mmHg for 30 minutes, despite anti-hypertensive therapy, within the past 24 hours)
   2. Coronary artery disease
   3. ST elevation myocardial infarction
   4. Acute coronary syndrome
   5. Hemodynamically significant dysrhythmia
   6. Congestive heart failure
   7. Cardiomyopathy (including Takotsubo cardiomyopathy)
   8. Other severe structural cardiac abnormalities
6. Renal

   a. Renal failure requiring renal replacement therapy (e.g. CVVH or HD)
7. Endocrine

   a. History of or clinical suspicion for thyrotoxicosis
8. Reproductive

   a. Pregnancy
9. Ophthalmologic

   a. History of glaucoma
10. Pharmacologic

    a. Monoamine oxidase inhibitor therapy within past 14 days
11. Other

    1. Any condition or finding that in the judgment of the PI or treating clinical team significantly increases the risk or significantly decreases the likelihood of a response to IV MPH

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2026-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Brian L Edlow, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Edlow BL, Barra ME, Zhou DW, Foulkes AS, Snider SB, Threlkeld ZD, Chakravarty S, Kirsch JE, Chan ST, Meisler SL, Bleck TP, Fins JJ, Giacino JT, Hochberg LR, Solt K, Brown EN, Bodien YG. Personalized Connectome Mapping to Guide Targeted Therapy and Promote Recovery of Consciousness in the Intensive Care Unit. Neurocrit Care. 2020 Oct;33(2):364-375. doi: 10.1007/s12028-020-01062-7. Epub 2020 Aug 13. PMID 32794142
- See also: Homepage of the Laboratory for NeuroImaging of Coma and Consciousness — https://www.comarecoverylab.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 10 patients were enrolled with informed consent provided by surrogate decision-makers, but one patient was withdrawn from the study by surrogate decision-makers prior to any study procedures were performed.
Period: Overall Study
Arm/Group | IV MPH
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: adults with severe TBI
Groups:
- IV MPH: 9 patients with severe traumatic brain injury (TBI), age range 25-77, all male.
Arm/Group | IV MPH
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (21.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 6
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events at Each Dose
Description: Adverse Events
  An AE is defined as any untoward medical occurrence associated with the use of an intervention in humans, whether or not considered intervention-related (21 CFR 312.32 (a)). In the STIMPACT Trial an AE may include, but is not limited to:
  * Sustained hypertension = SBP > 200 mmHg or DBP > 120 mmHg for > 30 min, refractory to medical therapy, or
  * Sustained tachycardia = HR > 120 bpm for > 30 min, refractory to medical therapy, or
  * Sustained intracranial hypertension = ICP > 25 mmHg for > 5 min, refractory to medical therapy
  Serious Adverse Events
  An AE or suspected adverse reaction is considered "serious" if, in the view of the investigator or the Independent Medical Monitor, it results in any of the following outcomes:
  * Death not related to withdrawal of life-sustaining therapy
  * A life-threatening event
  * Prolongation of existing hospitalization
  * Significant incapacity or substantial disruption of the ability to conduct normal life function
Time Frame: 4 Days
Population: 9 participants received the 0.5 mg/kg IV MPH dose and and the 1.0 mg/kg IV MPH dose. 6 participants received the 2.0 mg/kg IV MPH dose.
Measure: Count of Participants; unit: Participants
Groups:
- IV MPH: All patients received IV Methylphenidate (MPH). Patients received escalating daily doses of IV MPH starting at 0.5 mg/kg, increasing stepwise to 1.0mg/kg and 2.0 mg/kg unless an adverse event (AE) necessitated dose de-escalation or a serious adverse event (SAE) necessitated that the patient stop participation in the study.
Arm/Group | IV MPH
Number analyzed (Participants) | 9
Participants
  0.5 mg/kg IV MPH | 0
  1.0 mg/kg IV MPH | 2
  2.0 mg/kg IV MPH: number analyzed (Participants) | 6
  2.0 mg/kg IV MPH | 1

2. Secondary Outcome: Time to Maximal Serum Concentration of IV Methylphenidate (MPH)
Description: The median (range) time (hours) to maximum concentrations at 0.5, 1.0, and 2.0 mg/kg doses was measured.
Time Frame: 4 Days
Population: We measured the median (range) time (hours) to maximum concentrations at 0.5, 1.0, and 2.0 mg/kg doses of IV MPH.
Measure: Median (Full Range); unit: hours
Arm/Group | IV MPH
Number analyzed (Participants) | 9
hours
  0.5 mg/kg IV MPH | 0.12 [0.08 to 0.13]
  1.0 mg/kg IV MPH | 0.15 [0.07 to 0.18]
  2.0 mg/kg IV MPH: number analyzed (Participants) | 6
  2.0 mg/kg IV MPH | 0.23 [0.2 to 0.3]

3. Secondary Outcome: Serum Half-life of IV Methylphenidate (MPH)
Description: The mean (SD) serum half-lives (hours) at 0.5, 1.0, and 2.0 mg/kg doses was assessed.
Time Frame: 4 Days
Population: The mean (SD) serum half-lives (hours) at 0.5, 1.0, and 2.0 mg/kg doses was assessed.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | IV MPH
Number analyzed (Participants) | 9
hours
  0.5 mg/kg | 5.07 (2.55)
  1.0 mg/kg | 4.39 (1.92)
  2.0 mg/kg: number analyzed (Participants) | 6
  2.0 mg/kg | 5.01 (1.80)

4. Secondary Outcome: Cerebral Cortical Connectivity as Measured by fMRI
Description: We performed a change-point analysis of time-series resting-state fMRI data to determine if individual participants responded to the 2.0 mg/kg dose of IV MPH. Specifically, we measured resting-state fMRI connectivity between the brainstem ventral tegmental area and the default mode network after the bolus of IV MPH as compared to before the bolus of IV MPH. The bolus of IV MPH was administered in the MRI scanner while the patient was undergoing a 40-minute resting-state fMRI (10 minutes of data acquisition pre-bolus, 30 minutes of data acquisition post-bolus). The goal of the analysis was to determine if each patient responded to IV MPH, as defined by a positive change point (i.e., increase in connectivity after the bolus of IV MPH). Connectivity was measured via Pearson correlations using the software package CONN.
Time Frame: 4 Days
Population: Functional MRI data were obtained in two study participants.
Measure: Number; unit: number of responders
Arm/Group | IV MPH
Number analyzed (Participants) | 2
number of responders | 1

5. Secondary Outcome: Cerebral Cortical Connectivity as Measured by EEG
Description: We performed a change-point analysis of time-series resting-state EEG data to determine if individual participants responded to each dose of IV MPH. Specifically, we measured resting-state EEG background rhythm, using the alpha/delta ratio as a quantitative biomarker of overall brain function (i.e., alpha/delta ratio was measured for all EEG leads in a clinical 19-electrode montage). In a continuous time-series analysis of resting EEG data acquired 1 hour before and 1 hour after each IV MPH bolus, we tested for a "change-point" in the alpha/delta ratio, which represents a statistically significant increase in alpha/delta ratio. The goal of the analysis was to determine if each patient responded to IV MPH, as defined by a positive change point (i.e., increase in alpha/delta after the bolus of IV MPH). EEG analyses were performed using MATLAB software.
Time Frame: 4 Days
Population: EEG data were obtained in all nine study participants at the 0.5 mg/kg dose and 1.0 mg/kg dose, and in 6 participants at the 2.0 mg/kg dose.
Measure: Number; unit: number of responders
Arm/Group | IV MPH
Number analyzed (Participants) | 9
number of responders
  0.5 mg/kg IV MPH | 4
  1.0 mg/kg IV MPH | 2
  2.0 mg/kg IV MPH: number analyzed (Participants) | 6
  2.0 mg/kg IV MPH | 0

ADVERSE EVENTS:
Time Frame: 4 days
Groups:
- 0.5 mg/kg IV MPH: 9 patients received 0.5 mg/kg IV MPH.
- 1.0 mg/kg IV MPH: 9 patients received 1.0 mg/kg IV MPH.
- 2.0 mg/kg IV MPH: 6 patients received 0.5 mg/kg IV MPH.
Arm/Group | 0.5 mg/kg IV MPH | 1.0 mg/kg IV MPH | 2.0 mg/kg IV MPH
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/6
Other Adverse Events (participants affected / at risk) | 0/9 | 2/9 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.5 mg/kg IV MPH (N=9) | 1.0 mg/kg IV MPH (N=9) | 2.0 mg/kg IV MPH (N=6)
Paroxysmal Sympathetic Hyperactivity (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — assessed at bedside in ICU
Insomnia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — assessed at bedside in ICU
Emesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — assessed at bedside in ICU
Transaminitis (increased ALT/AST) (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) — assessed via lab analysis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-16): https://cdn.clinicaltrials.gov/large-docs/56/NCT03814356/Prot_SAP_000.pdf